CLINICAL TRIAL: NCT00802789
Title: Montelukast in Chronic Asthma: Non-interventional Study With Montelukast 10 mg
Brief Title: Montelukast in Chronic Asthma
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0476-421; 2008_031 (Other: Merck); MK-0476-421
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Mild to moderate adult asthmatics (≥18years of age) insufficiently treated with ICS or ICS + LABA.

SUMMARY:
Treatment of patients insufficiently treated with ICS or ICS + LABA.

ELIGIBILITY:
Inclusion Criteria:

* Patients Insufficiently Treated With ICS Or ICS + LABA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mild to moderate adult asthmatics (≥18 years of age) insufficiently treated with ICS or ICS + LABA
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2007-04; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Documentation of asthma control via ACT (Asthma Control Test). | 6 months (12 months optional)

SECONDARY OUTCOMES:
Mini Asthma Quality of Life Questionnaire (Mini AQLQ). | 6 months (12 months optional)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Virchow JC, Mehta A, Ljungblad L, Mitfessel H; MONICA study group. Add-on montelukast in inadequately controlled asthma patients in a 6-month open-label study: the MONtelukast In Chronic Asthma (MONICA) study. Respir Med. 2010 May;104(5):644-51. doi: 10.1016/j.rmed.2009.11.022. Epub 2009 Dec 23. PMID 20031382